CLINICAL TRIAL: NCT04241328
Title: SYMBIOSIS Post-Market Registry
Brief Title: Medtronic SYMBIOSIS Post-Market Registry for Patients Undergoing Cardiac Surgery
Acronym: SYMBIOSIS
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT19022PMF001
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational, multi-center prospective, post-market registry is to confirm real-world device safety and performance, to ensure the continued acceptability of identified risks, and detect emerging risks.

DETAILED DESCRIPTION:
The objective is to collect product safety and performance data for Medtronic CE (Conformitè Europëenne )-Marked Cardiac Surgery, including perfusion (CS) products.

The main goals of this data collection are as follows:

* Identification of any (new) device-related complications including events which were not anticipated or documented in the Instructions For Use (IFU), or Risk Management Plan, or Clinical Evidence Evaluation report, or Design Failure Modes and Effect Analysis
* Evaluation of device success defined as the absence of any probable or causal device-related adverse events or device deficiencies
* Evaluation of general device performance when applicable

Subjects are enrolled and, if applicable, followed according to routine care practices at their treating hospital.

Inclusion Criteria:

* Subject or legally authorized representative provides written data release and/or informed consent per institution and/or geographical requirements prior to discharge from participating Registry hospital.
* Subject will undergo or underwent a procedure in which an eligible Medtronic CS product is/was used.

Exclusion Criteria:

• Currently participating in an interventional drug or device study which may induce confounding factor(s) to the results from this Registry

Data collection includes, for example:

* Demographics
* Product performance information
* Safety Events

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative provides written data release and/or informed consent per institution and/or geographical requirements prior to discharge from participating registry hospital.
* Subject will undergo or underwent a procedure in which an eligible Medtronic CS product is/was used.

Exclusion Criteria:

* Currently participating in an interventional drug or device study which may induce confounding factor(s) to the results from this Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive subjects with the intent of being treated or treated (up to discharge from treating hospital) with a market-approved Medtronic CS product, are candidates to be enrolled. The Investigator will determine subject eligibility in SYMBIOSIS based upon the inclusion/exclusion criteria. If a subject meets all inclusion and none of the exclusion criteria, they will be informed about the SYMBIOSIS Registry. SYMBIOSIS will collect data of numerous patient conditions for which Medtronic CS products are being used.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Safety | Procedural
  Procedure- , device-related events and device deficiencies
Device performance | Procedural
  Device Success

CONTACTS AND LOCATIONS:
Locations (14):
- AKH Wien, Vienna, Austria
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven, Leuven
- France (2):
  - CHU d'Angers, Angers
  - Clinique Claude Bernard, Metz
- Germany (3):
  - Uniklinik RWTH Aachen, Aachen
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum München, Munich
- Onassis Hospital, Athens, Greece
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht University Medical Center (MUMC+), Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
- Haukeland Universitetssjukehus, Bergen, Norway
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No